CLINICAL TRIAL: NCT06389305
Title: Cytokine-induced Killer(CIK) Cell Therapy and Its Impact on Early Functional Exhaustion of Chimeric Antigen Receptor-T(CAR-T) Cells in Relapsed or Refractory Acute B-Lymphoblastic Leukemia: A Prospective Study
Brief Title: CIK Cell Therapy for Relapsed or Refractory Acute B-Lymphoblastic Leukemia: Prognostic Impact on Patients With Early CAR-T Cell Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2024-012
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia, in Relapse; Refractory Acute Lymphoid Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: a prospective cohort study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peripheral blood lymphocytes (Placebo Comparator)
  Interventions: Drug: peripheral blood lymphocytes
- CIK cells (Experimental)
  Interventions: Drug: CIK cell

INTERVENTIONS:
Drug: peripheral blood lymphocytes — autologous or allogeneic peripheral blood lymphocytes
  Arms: peripheral blood lymphocytes
Drug: CIK cell — autologous or allogeneic cytokine-induced killer (CIK) cells
  Arms: CIK cells

SUMMARY:
This is a single-center, double-blind, randomized trial. Patients with relapsed or refractory acute B-lymphoblastic leukemia(r/r B-ALL) experiencing early functional exhaustion of CAR-T cells will be randomly allocated into three groups: the control cell group, the CIK treatment group, and the messenger RNA(mRNA)-CIK treatment group. The primary objective of the study is to evaluate the prognostic impact of CIK cell therapy on the early functional exhaustion of CAR-T cells in children and adolescent and young adult (AYA) with r/r B-ALL. The primary endpoint of the study is the event-free survival rate of these patient in the CIK cell therapy group.A total number of 213 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* A patient must meet all of the following to be enrolled:

  1. A confirmed diagnosis of refractory or relapsed B-ALL (criteria reference: NCCN, 2024.4), where all patients meet the National Comprehensive Cancer Network(NCCN) guidelines for the diagnosis of acute lymphoblastic leukemia (hematopathological examination of bone marrow aspirate and biopsy tissue showing ≥20% lymphoblasts in the bone marrow, confirmed by comprehensive flow cytometry (FCM) immunotyping, minimal residual disease analysis, and G-banded metaphase chromosome karyotype analysis). Molecular characteristics can be described through methods such as interphase fluorescence in situ hybridization (FISH) testing, reverse transcription polymerase chain reaction (RT-PCR) testing, and next-generation sequencing (NGS) for comprehensive detection of fusion genes and pathogenic mutations. Determination can also be made by the World Health Organization's subtypes of acute lymphoblastic leukemia, as well as cytogenetic and clinical risk groups.
  2. Loss of CAR-T cell activity within 6 months after previous CAR-T therapy and no relapse.
  3. Age between 1 and 39 years old.
  4. No severe allergic constitution.
  5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
  6. Life expectancy, as judged by the investigator, of at least 60 days.
  7. Patients with self-awareness between 8 and 39 years of age voluntarily sign an informed consent, and the legal representative (guardians) of child patients under 18 years of age voluntarily signs an informed consent.

Exclusion Criteria:

* A patient with at least one of the following conditions will be excluded:

  1. Received bendamustine treatment within the past 9 months;
  2. Intracranial hypertension or impaired consciousness in the brain;
  3. Symptomatic heart failure or severe arrhythmia;
  4. Symptoms of severe respiratory failure;
  5. With other types of malignant tumors;
  6. Disseminated intravascular coagulation;
  7. Serum creatinine and/or blood urea nitrogen ≥ 1.5 times the normal value;
  8. Suffering from sepsis or other uncontrollable infections;
  9. Uncontrollable diabetes;
  10. Severe mental disorders;
  11. Significant lesions in the brain as detected by head magnetic resonance imaging;
  12. Leukemic cells in the cerebrospinal fluid >20 cells/μL;
  13. Peripheral blood leukemic cell proportion >30%;
  14. Have undergone organ transplantation;
  15. Female patients (those with childbearing potential) are pregnant or lactating;
  16. Active or uncontrollable infectious diseases, such as hepatitis (HBV, HCV), HIV, or syphilis.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 213 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival(EFS) in CIK infusion group | 2-year EFS rate
  EFS is defined as the time from CIK-cell infusion to the earliest relapse, death from any cause, or treatment failure

SECONDARY OUTCOMES:
Progression-free survival(PFS) in CIK infusion group | 2-year PFS rate
  PFS is defined as the time from CIK-cell infusion until objective tumor progression or death depending on study protocol
Duration of response(DOR) in CIK infusion group | from enrollment to the end of treatment at 15 years
  DOR is defined as the time interval from the earliest qualifying minimal residual disease-negative response [i.e. complete remission(CR),complete remission with partial hematological recovery(CRh), complete remission with incomplete hematological recovery(CRi), morphologic leukemia-free state(MLFS), or aplastic marrow (patients with blood and bone marrow disease), central nervous system(CNS) remission (patients with CNS disease) and complete resolution of the lymphomatous enlargement by CT or positron emission tomography(PET)-CT negative (for patients with a previous positive PET-CT) (patients with lymphomatous extramedullary disease)] to the date of relapse or death from any cause.
Overall survival(OS) in CIK infusion group | from enrollment to the end of treatment at 15 years
  OS is defined as the time from CIK-cell infusion to death from any cause.
EFS in mRNA-CIK infusion group | 2-year EFS rate
  EFS is defined as the time from mRNA-CIK-cell infusion to the earliest relapse, death from any cause, or treatment failure

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No